CLINICAL TRIAL: NCT01009866
Title: Phase I Study of Immunotoxin, MR1-1
Brief Title: Study of Immunotoxin, MR1-1
Acronym: MR1-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Darell D. Bigner, MD, PhD (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Darell D. Bigner, MD, PhD, Director, The Preston Robert Tisch Brain Tumor Center at Duke, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011617; P50NS020023 (NIH)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Supratentorial Malignant Brain Tumor
Keywords: Malignant brain tumor; GBM; recurrent brain tumor; Supratentorial malignant brain tumor; astrocytomas; ependymomas; Residual, progressive, or recurrent supratentorial malignant brain tumor based on imaging studies with measurable; disease (>0.5cm).
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Ependymoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR1-1 (Experimental): All subjects are enrolled onto this arm. All subjects will receive MR1-1.
  Interventions: Biological: MR1-1

INTERVENTIONS:
Biological: MR1-1 — Based on preclinical toxicity studies, the starting total drug dose will be 0.5μg (500ng) which represents 1/20th of the MTD in rats. The infusion flow rate will be fixed at 0.5 mL/h from each of two catheters. A total of 96 mLs of drug solution will be delivered over 96 hours. MR1-1KDEL dose escalation will be accomplished by increasing drug concentration allowing flow rate and infusion volume to remain unchanged. Drug dose will be doubled in successive cohorts so long as DLTs are not observed as follows: 25 ng/mL (2.4 μg)(starting dose); 50ng/mL (4.8μg); 100 ng/mL (9.6μg); 200ng/mL (19.2μg); 400 ng/mL (38.4μg); 800 ng/mL (76.8μg); and 1600 ng/mL (153.6μg).
  Other Names: MR1-1KDEL

SUMMARY:
Purpose of the study:

Primary Objective: Determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of MR1-1KDEL when delivered intracerebrally by convection-enhanced delivery (CED) in patients with supratentorial malignant brain tumors.

Secondary Objective: Document any radiographic responses associated with intracerebral CED of MR1-1KDEL.

Hypothesis: The investigators believe that MR1-1KDEL will be an effective anti-tumor agent for patients with supratentorial malignant brain tumors when delivered by CED.

Design & procedures: This protocol is designed primarily to determine the MTD and DLT of a novel, tumor-specific immunotoxin, MR1-1KDEL. MR1-1KDEL will be delivered intracerebrally by CED using 2 intracerebral catheters with at least one catheter placed within the enhancing portion of the tumor. 124I-labeled albumin will be co-infused with gadolinium and PET and MRI images will be obtained at the conclusion of the infusion to monitor volume of drug distribution and leakage into the CSF space.

Based on preclinical toxicity studies, the starting total drug dose will be 0.5μg (500ng) which represents 1/20th of the MTD in rats. The infusion flow rate will be fixed at 0.5 mL/h from each of two to four catheters. A total of 144 mLs of drug solution will be delivered over 72 hours. MR1-1KDEL dose escalation will be accomplished by increasing drug concentration allowing flow rate and infusion volume to remain unchanged. Drug dose will be doubled in successive cohorts so long as DLTs are not observed as follows: 25 ng/mL (2.4 μg)(starting dose); 50ng/mL (4.8μg); 100 ng/mL (9.6μg); 200ng/mL (19.2μg); 400 ng/mL (38.4μg); 800 ng/mL (76.8μg); and 1600 ng/mL (153.6μg). At least 3 patients will be enrolled in each cohort. All patients in a given cohort will be observed for at least two weeks following infusion of the study drug before patients in the next cohort are treated. If no patients in a given cohort experience a DLT, the dose will be escalated in the next cohort. If 1 out of 3 patients in a given cohort experience DLT, 3 additional patients will be entered in that cohort. If 2 patients develop a DLT in any cohort of 3 or 6 patients, the previous dose will be declared the MTD. Patients will be followed at 1, 3, 6, 9, 12 month intervals for toxicity and adverse events, radiographic response, and survival. Patients will be off study when progressive disease is documented.

Risk/benefit assessment: This is an experimental study and unforeseeable or unexpected risks may be involved.

ELIGIBILITY:
Inclusion Criteria:

* Residual, progressive, or recurrent supratentorial malignant brain tumor based on imaging studies with measurable disease (>0.5cm).
* Patient will have completed some form of radiation therapy prior to toxin treatment.
* Karnofsky Performance score >70.
* The presence of the target antigen, EGFRvIII, must be identified on tumor tissue by immunohistochemistry.
* Platelet count > 100 x 109/L; PTT and PT < 120% of normal range.
* Creatinine < 120% of normal range.
* Total bilirubin, SGOT, SGPT,alkaline phosphatase < 300% of normal range.

Exclusion Criteria:

* Patients who are pregnant, breast-feeding, or unwilling to practice an effective method of birth control.
* Patients with known potentially anaphylactic allergic reactions to iodine or gadolinium-DTPA.
* Patients who cannot undergo MRI due to obesity or to having certain metal in their bodies (specifically pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods or plates).
* Patients that have not recovered from the toxic effects of prior chemotherapy and/or radiation therapy.
* Patients with an impending, life-threatening cerebral herniation syndrome.
* Patients with subependymal or CSF disease.
* Patients who are under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose limiting toxicity | continual

SECONDARY OUTCOMES:
Disease Progression | continual

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States